CLINICAL TRIAL: NCT06456164
Title: IntraCERvical Balloon Catheter in the Setting of Induction of Labor for Fetal Loss or Abortion (CERBI): a Pilot Randomized Controlled Trial
Brief Title: IntraCERvical Balloon Catheter in the Setting of Induction of Labor for Fetal Loss or Abortion
Acronym: CERBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has not received IRB approval.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB24-0835
Record Dates: First submitted 2024-05-19; First posted 2024-06-13 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Abortion, Complete; Fetal Death; Induction of Labor Affected Fetus / Newborn
Keywords: induction termination; medication abortion
MeSH Terms: conditions — Fetal Death

STUDY DESIGN:
Intervention Model Description: Cook Cervical Ripening Balloon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Usual Care (No Intervention): Participants will receive mifepristone 200 mg by mouth 24 hours prior to induction of labor. Labor will be induced with use of vaginal misoprostol according to regimens endorsed by the American College of Obstetricians and Gynecologists and the Society of Family Planning.
- Usual care with mechanical dilation (Experimental): Participants will receive mifepristone 200 mg by mouth 24 hours prior to induction of labor. Participants will have their labor induced concomitantly with misoprostol (according to the regimen described in the "Usual Care" arm) and placement of the Cook Cervical Ripening Balloon.
  Interventions: Device: Cook Cervical Ripening Balloon

INTERVENTIONS:
Device: Cook Cervical Ripening Balloon — The Cook Cervical Ripening Balloon is a double-balloon catheter designed to mechanically ripen the cervix prior to labor induction when the cervix is unfavorable for induction.
  Arms: Usual care with mechanical dilation

SUMMARY:
The goal of this research is to understand whether it is practical and safe to use an intracervical balloon catheter in addition to standard of care medications at the time of an induction of labor for an abortion or fetal death. The medical device used in this study is cleared by the Food and Drug Administration (FDA) and is used for induction of labor at term gestational ages (at or above 37 weeks of gestation). The study team will also collect data about patient-level experiences with the procedure, time in labor, and labor-related complications, such as higher-than-expected blood loss or infection.

DETAILED DESCRIPTION:
Commonly, induction of labor in the second trimester is accomplished with the use of oral anti-progestin medications (i.e., mifepristone) at least 24 hours prior to administration of sublingual, buccal, or vaginal prostaglandins (e.g., misoprostol). Innovation over the past decade has largely been focused on the concomitant use of mechanical dilation for induction of labor in order to reduce the time from initiation of labor to delivery. However, limited data exist to demonstrate the efficacy of an intracervical balloon catheter during second-trimester induction of labor. Therefore, the principal investigator seeks to conduct a feasibility randomized controlled trial to evaluate whether an intracervical balloon catheter - commonly used for inductions of labor at later gestational ages - can be used during second-trimester inductions of labor.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18
* English or Spanish-speaking
* Cervical dilation < 3 centimeters
* Gestational age between 22w0d and 27w6d

Exclusion Criteria:

* Maternal age < 18
* Non-English- or Spanish-speaking
* Cervical dilation ≥ 3 centimeters
* Gestational age below 22w0d or above 27w6d
* Allergy to mifepristone or misoprostol
* Hemolysis, Elevated Liver Enzymes, and Low Platelets (HELLP) syndrome
* Disseminated intravascular coagulopathy
* Placenta previa or suspected placenta accreta spectrum disorder
* Placental abruption
* Suspected intraamniotic infection
* Rupture of membranes
* Untreated genitourinary tract infection
* 3 or more cesarean deliveries, classical cesarean delivery, or endometrial cavity-entering myomectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants diagnosed with clinical chorioamnionitis or postpartum endometritis | Up to 6 weeks post-delivery
  Maternal temperature greater than 39°C or 38-38.9°C with evidence of leukocytosis or purulent cervical drainage
Number of participants diagnosed with sepsis | Up to 6 weeks post-delivery
  Sepsis in Obstetrics Score > 6. Score calculated from maximum maternal temperature, blood pressure, heart rate, respiratory rate, oxygen saturation, white blood cell count, and serum lactic acid
Number of participants diagnosed with septic shock | Up to 6 weeks post-delivery
  Hypotension requiring vasopressors to maintain mean arterial pressure ≥65 mm Hg and serum lactate level >2 mmol/L (18mg/dL) despite adequate volume resuscitation
Number of participants diagnosed with postpartum hemorrhage | Up to 6 weeks post-delivery
  Estimated or quantitative blood loss greater than 1000 mL at the conclusion of expulsion of the fetus and placenta
Number of participants requiring blood transfusion after expulsion of the fetus and placenta | Up to 6 weeks post-delivery
Number of participants requiring uterotonics | Up to 6 weeks post-delivery
  Need for misoprostol, carboprost, and/or methergine after expulsion of the fetus and/or placenta
Number of participants diagnosed with a cervical laceration | During delivery hospitalization (within 72 hours after delivery)
Number of participants requiring adjunctive procedures in the setting of postpartum hemorrhage | Up to 6 weeks post-delivery
  Dilation and curettage, insertion of intrauterine tamponade device (i.e., Bakri or Jada devices), uterine artery embolization, exploratory laparotomy, O'Leary and/or B-Lynch sutures, and/or other uterine-conserving surgical measures to control hemorrhage
Number of participants requiring hysterotomy or dilation and evacuation | During delivery hospitalization (within the first 72 hours after admission)
  Need for hysterotomy or dilation and evacuation in setting of failed induction of labor
Number of participants diagnosed with a uterine rupture | Within the first 12 hours after expulsion of the fetus
Number of participants requiring intensive care unit admission | Up to 6 weeks post-delivery
Number of participants requiring readmission to the hospital within 6 weeks of delivery | Up to 6 weeks post-delivery
Number of participants who experience death | Up to 6 weeks post-delivery

SECONDARY OUTCOMES:
Patient-reported pain | Up to 6 weeks post-delivery
  Use of visual analog scale (0-10), with higher scores indicating worse levels of pain
Patient-reported distress | Up to 6 weeks post-delivery
  Impact of Event scale (0-88), with higher scores indicating higher levels of distress
Patient-reported acceptability of intervention | Up to 6 weeks post-delivery
  assessed via the question "Would you have the same procedure again if you had to have another second-trimester induction of labor?" and "Did you think the second-trimester induction of labor was better or worse than expected?"
Patient-reported satisfaction | During intrapartum period (up to 72 hours after delivery)
  Client Satisfaction Questionnaire-8 (8-22), with higher scores indicating higher levels of satisfaction
Total duration of labor, in hours | During intrapartum period (up to 72 hours after delivery)
  Total duration from initiation of misoprostol to expulsion of the fetus, in hours
Total blood loss, in milliliters | Within the first 24 hours after expulsion of the fetus and placenta
  Total blood loss after expulsion of the fetus and placenta
Number of participants requiring dilation and curettage or manual extraction of the placenta | Within the first 12 hours after expulsion of the fetus

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Premkumar, MD PhD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: Yes
Once data are peer-reviewed and published, the investigators will plan to share individual participant data with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 1 year after completion of data analysis,